CLINICAL TRIAL: NCT06775782
Title: Remote Ischemic Conditioning for Acute Moderate Ischemic Stroke Due to Large Artery Atherosclerosis: A Multi-centered, Open-label, Blind Endpoint, Randomized Controlled Trial
Brief Title: Remote Ischemic Conditioning for Acute Moderate Ischemic Stroke Due to Large Artery Atherosclerosis
Acronym: RIC-LAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2023-003
Record Dates: First submitted 2025-01-08; First posted 2025-01-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke；Large Artery Atherosclerosis；Remote Ischemic Conditioning therapy; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke | interventions — Therapeutics; Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning + Medical Management (Experimental): Patients in this group will receive Remote Ischemic Conditioning plus best medical management.
  Interventions: Device: Remote Ischemic Conditioning (RIC) treatment; Drug: Medical Management
- Medical Management (Active Comparator): Patients in this group will receive best medical management alone.
  Interventions: Drug: Medical Management

INTERVENTIONS:
Device: Remote Ischemic Conditioning (RIC) treatment — RIC will be given twice a day for 10-14 days. RIC will be applied using an automated RIC device. The cuff of the RIC medical device will be placed around the bilateral upper limbs. Five cycles of cuff inflation (200mmHg for 5 minutes) and deflation (for 5 minutes) for a total procedure time of 50 minutes.
  Arms: Remote Ischemic Conditioning + Medical Management
Drug: Medical Management — Patients will receive standard guideline-directed medical therapy, which will include monitor vital signs, management of blood pressure, glucose and lipids, antithrombotic therapy if appropriate.

SUMMARY:
Large Artery Atherosclerosis is one of the most prevalent causes of stroke worldwide and is associated with a high risk of disability and recurrent strokes. Remote Ischemic Conditioning (RIC) is a promising therapy, and it has been recommended for further investigation in patients with acute ischemic stroke resulting from large artery atherosclerosis. The primary objective of this study is to assess the efficacy of RIC in patients suffering from acute moderate ischemic stroke due to large artery atherosclerosis.

DETAILED DESCRIPTION:
This multi-centered, open-label, blind endpoint, randomized controlled trial aims to investigate the efficacy of RIC in patients with acute moderate ischemic stroke due to large artery atherosclerosis. A total of 1150 participants (age 18 to 85 years) within 48 hours of symptom onset of acute moderate ischemic stroke (NIHSS score 6-16, or NIHSS score 4-5 with disabling deficits) due to large artery atherosclerosis will be enrolled. Eligible patients will be randomized in a 1:1 ratio into RIC treatment plus medical management versus medical management alone after offering informed consent.

The primary endpoint is excellent functional outcome at 90 days, defined as a modified Rankin Scale score of 0 to 1, which will be evaluated by independent researchers in the blind state.

ELIGIBILITY:
Inclusion Criteria

1. Male or female with age from 18 to 85 years old;
2. Randomization must be within 48 hours after stroke symptom onset;
3. Ischemic stroke confirmed by MRI diffusion-weighted imaging;
4. NIHSS score 6-16, or 4-5 with disabling deficits at the time of randomization. The following typically should be considered disabling deficits: Complete hemianopsia (≥2 on NIHSS question 3) or severe aphasia (≥2 on NIHSS question 9), or visual or sensory extinction (≥1 on NIHSS question 11) or any weakness limiting sustained effort against gravity (≥2 on NIHSS question 6 or 7);
5. Proven large vessel 50%-99% stenosis or occlusion by MRA, CTA or DSA in cervical or intracranial carotid artery, M1 or M2 segments of the middle cerebral artery, A1 segment of anterior cerebral artery, P1 segment of posterior cerebral artery, vertebral artery, or basilar artery. For patients with single cerebral infarction, when MRA indicates >50% stenosis rather than occlusion, CTA or DSA should be performed to exclude the risk of MRA overestimating stenosis severity. Acute neurological deficit and cerebral infarction are compatible with ischemia in the vascular territory;
6. Pre-stroke modified Rankin Scale score (mRS) of 0-1;
7. Signed Informed Consent obtained.

Exclusion Criteria

1. Thrombolysis or endovascular therapy performed or planned for index event;
2. Suspected or confirmed cardioembolic source of stroke: i. The aetiology of cardiogenic embolism with high embolic potential, such as atrial fibrillation, atrial flutter, rheumatic mitral or aortic stenosis, artificial heart valve, left atrial myxoma, valve neoplasm, left ventricular wall thrombus, congestive heart failure, bacterial endocarditis, cardiomyopathy, myocardial infarction within previous 30 days; ii. Multiple cerebral infarctions in more than one vascular territory (e.g., bilateral MCA, or an MCA and a basilar artery) confirmed MRI diffusion-weighted imaging;
3. Suspected or confirmed uncommon causes of cerebrovascular disorders: arterial dissection, Moyamoya disease, vasculitis disease, neurosyphilis, radiation induced vasculopathy, fibromuscular dysplasia, benign angiopathy of central nervous system, post-partum angiopathy, suspected vasospastic process, suspected recanalized embolus etc.;
4. Subclavian artery stenosis ≥ 50% or subclavian steal syndrome;
5. Refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg after drug treatment);
6. Evidence of intracranial tumor (except small meningioma), abscess, arteriovenous malformation;
7. Patients with bleeding propensity: platelet count <50×10^9/L; heparin was administered within 48 hours with APTT≥35s; on anticoagulant therapy with warfarin and International Normalized Ratio (INR) > 1.7;
8. Undergoing hemodialysis or peritoneal dialysis, or known severe renal insufficiency with glomerular filtration rate <30 ml/min or serum creatinine >220 mmol/L (2.5mg/dl);
9. Respiratory failure, including type I and type II;
10. Any contraindication for Remote Ischemic Conditioning: severe soft tissue injury, fracture, peripheral vascular disease, arteriovenous fistula, or venous thrombosis in the upper limbs;
11. Severe comorbid condition with life expectancy < 6 months；
12. Current participation in any other investigational trial；
13. Pregnancy；
14. Patients not suitable for this clinical study considered by researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) 0-1 at 90 days | at 90 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of patients who have suffered from a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms. Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) 0-2 at 90 days | at 90 days after randomization
Distribution of the Modified Rankin Scale (mRS) at 90 days | at 90 days after randomization
Early neurological deterioration within 48 hours | within 48 hours after randomization
Change of NIHSS scores from baseline to 12 days | at 12 days after randomization
Recurrence of Ischemic stroke within 90 days | within 90 days after randomization
Quality of life measured by Euro-QoL-5D-5L at 90 days | at 90 days after randomization
Death due to any cause within 90 days | within 90 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No